CLINICAL TRIAL: NCT02406287
Title: A Controlled Study of the Aqueous Humor Dynamics of AR-13324 Ophthalmic Solution in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS102
Record Dates: First submitted 2015-03-12; First posted 2015-04-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — netarsudil; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Netarsudil (AR-13324) Ophthalmic Solution
  Interventions: Drug: Netarsudil (AR-13324) Ophthalmic Solution
- Placebo (Placebo Comparator): Netarsudil (AR-13324) Ophthalmic Solution Placebo
  Interventions: Drug: Netarsudil (AR-13324) Ophthalmic Solution Placebo

INTERVENTIONS:
Drug: Netarsudil (AR-13324) Ophthalmic Solution — Topical ophthalmic solution
  Arms: Active
Drug: Netarsudil (AR-13324) Ophthalmic Solution Placebo — Ophthalmic solution once a day
  Arms: Placebo

SUMMARY:
To evaluate the effect of netarsudil (AR-13324) ophthalmic solution on aqueous humor dynamics relative to its placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects at least 18 years of age.
2. Local area resident, existing patient or employee of Mayo Clinic.
3. Medically healthy subjects with clinically insignificant screening results.
4. Subjects with two normal (non-diseased) eyes.
5. Intraocular pressure between 14 and 21 mm Hg (inclusive) in each eye at screening.
6. Best-corrected visual acuity in each eye of +0.4 (20/50) or better.
7. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

1. Chronic or acute ophthalmic disease including glaucoma, macular degeneration, uveitis clinically significant cataract.
2. Known hypersensitivity to any component of the formulation or to topical anesthetics.
3. Previous intraocular surgery, retina laser procedures or refractive surgery.
4. Myopia greater than -4.00 D spherical equivalent.
5. Hyperopia greater than +2.00 D spherical equivalent.
6. Ocular trauma within the past six months.
7. Evidence of ocular infection, inflammation, cystoid macular edema, clinically significant blepharitis or conjunctivitis, or a history of herpes simplex keratitis.
8. Ocular medication of any kind within 30 days of screening.
9. Any abnormality preventing reliable applanation tonometry of either eye.
10. Central corneal thickness less than 500 μm or greater than 600 μm.
11. Cannot demonstrate proper delivery of the eye drop.
12. Clinically significant systemic disease which might interfere with the study.
13. Participation in any investigational study within the past 30 days prior to screening.
14. Use of systemic medication that could have a substantial effect on intraocular pressure within 30 days prior to screening, or anticipated during the study.
15. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a physician-supervised form of birth control for at least the last 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in aqueous humor flow rate measured by non-contact fluorophotometer | Day 1 compared to Day 8
  Aqueous humor flow rate measured by non-contact fluorophotometer; change from baseline
Change in outflow facility measured non-invasively by tonography | Day 1 compared to Day 8
  Outflow facility measured non-invasively by tonography; change from baseline
Change in episcleral venous pressure measured non-invasively by slit-lamp exam | Day 1 compared toDay 8
  Episcleral venous pressure measured non-invasively by slit-lamp exam; change from baseline
Change in visual acuity measured using eye chart | Day 1 compared to Day 8
  Visual acuity measured using eye chart; change from baseline
Change in biomicroscopy exam using non-invasive slit-lamp to evaluate cornea, conjunctiva, and anterior chamber of eye | Day 1 compared to Day 8
  Biomicroscopy exam using non-invasive slit-lamp to evaluate cornea, conjunctiva, and anterior chamber of eye; change from baseline

SECONDARY OUTCOMES:
Safety - Number of participants with adverse events | Day 1 compared to Day 8
  Number of participants with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ramirez, Study Director — Aerie Pharmaceuticals
Locations (1):
- Aerie Pharmaceutical, Bedminster, New Jersey, United States